CLINICAL TRIAL: NCT06866379
Title: Involvement of the Septal Nuclei of the Human Brain in Alcohol Use Disorder - a Functional Magnetic Resonance Imaging Study
Brief Title: Involvement of the Septal Nuclei of the Human Brain in Alcohol Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anders Fink-Jensen, MD, DMSci (Other)
Collaborators: Neurobiology Research Unit, Rigshospitalet (Unknown); The foundation of Mr. Ivan Nielsen (Unknown); King Christian X foundation (Unknown)
Responsible Party: Sponsor-Investigator, Anders Fink-Jensen, MD, DMSci, Professor, Senior Consultant, dr.med., Psychiatric Centre Rigshospitalet
Organization: Psychiatric Centre Rigshospitalet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: The septum study
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol use disorder; AUD; septum; fMRI; Brain imaging
MeSH Terms: conditions — Alcoholism | interventions — Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with AUD (Experimental): Participants diagnosed with alcohol use disorder participating in one fMRI brain scan.
  Interventions: Other: Brain imaging

INTERVENTIONS:
Other: Brain imaging — fMRI session with the ALCUE paradigme.

SUMMARY:
Alcohol activates reward systems in different brain areas, i.e., the nucleus accumbens, dorsal striatum, extended amygdala, and prefrontal cortex. These areas are all part of the reward neurocircuitry, which plays an important role in the development of addiction.

A former study performed on rodents has shown that a specific area of the forebrain, the septal nuclei, is associated with the feeling of reward and, hence, addiction when stimulated. However, whether the septal area is involved in reward and addiction in humans is sparsely investigated.

The purpose of this brain-imaging study is to assess how the septal nuclei react to alcohol-related pictures shown to participants diagnosed with alcohol use disorder while lying in an MRI scanner, compared to people without a diagnosis of alcohol use disorder. This might give us a better understanding of how the septal nuclei is involved in reward and addiction.

DETAILED DESCRIPTION:
This is a comparative, non-interventional, case-control, brain imaging study using the ALCUE paradigm to investigate the neuro-anatomical underpinings of AUD during a fMRI-scan. The contrast used for the fMRI scans is the BOLD signal which measures the ratio of oxygenated to deoxygenated blood in the brain as a measurement of neural activity.

The study will conclude after the last participant with AUD succesfully has undergone the fMRI scan, and will include 50 participants in total: 25 participants diagnosed with AUD and 25 participants without AUD (data from a previous brain imaging study). Written informed consent will be collected, before any trial activities are performed.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with alcohol use disorder (AUD) according to DSM-5, and alcohol dependence according to ICD-10
* An Alcohol Use Disorder Identification Test (AUDIT) score ≥ 15
* At least six heavy drinking days for the last 30 days, measured with the Time Line Follow Back (TLFB) method

Exclusion criteria:

* Diagnosis of schizophrenia spectrum disorder, paranoid psychosis, bipolar disorder, or mental retardation
* Previous or current substance use disorder other than AUD and nicotine use disorder
* History of alcohol withdrawal seizures within the past 5 years
* Alcohol withdrawal symptoms defined as a CIWA-Ar score > 9 at screening or at the fMRI session
* Treatment with chlordiazepoxide or other benzodiazepine within the past 30 days
* Other pharmacological treatment for AUD within the past 30 days
* Treatment with GLP-1 analogues within the last 6 months
* Urine tests positive for psychoactive drugs (cocaine, amphetamine, TCH, methadone, opioids, and benzodiazepines) at screening
* DUDIT score ≥ 2/6 for females/males
* Contraindications for undergoing an fMRI scan (magnetic implants, metal splinters, pacemaker, claustrophobia, etc.)
* Females of childbearing potential who are either pregnant, breastfeeding or have the intention of becoming pregnant within the next month or are not using contraception appropriate for participating in a clinical study
* Pregnancy (positive urine pregnancy test)
* Unable to speak or understand Danish
* Any condition that the investigator feels would interfere with trial participation

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Significant differences in alcohol cue related fMRI BOLD signals in the septal nuclei of the brain between AUD patients and healthy controls. | 12 minutes while the brain scan is being conducted
  Data is obtained using the ALCUE fMRI paradigm with the septal area as a predefined region of interest (ROI).

SECONDARY OUTCOMES:
Significant differences between AUD patients and healthy controls with respect to the subjectively reported craving degree | From beginning of the fMRI scan to the end of it at 12 minutes
  The craving degree will be measured during the fMRI paradigm on a visual analogue scale ranging from 0 (no craving) to 100 (extremely extensive craving)
Significant differences between AUD patients and healthy controls with respect to alcohol cue related signals | From beginning of the fMRI scan to the end of it at 12 minutes
  The differences will be measured during the fMRI scan and analysed with BOLD-respons in putamen, caudate, nucleus accumbens and dorsal- and ventral striatum.
Correlation between subjectively reported craving and BOLD signals | From beginning of the fMRI scan to the end of it at 12 minutes
  A comparision between the subjectively measured craving degree using a visual analogue scale and the BOLD signals of the putamen, caudate, nucleus accumbens and dorsal- and ventral striatum measured during the fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Center Copenhagen, Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided